CLINICAL TRIAL: NCT05670769
Title: The Effect of Home Midwifery Care Given to Pregnant Women Diagnosed With Gestational Diabetes on Attitudes and Self-Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cemile Onat Koroglu, Lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 04.11.2022/37
Record Dates: First submitted 2022-12-20; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Gestational Diabetes; Pregnancy, High Risk
Keywords: Midwifery; home care; gestational diabetes; attitude, self care
MeSH Terms: conditions — Diabetes, Gestational; Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): * All forms will be filled in by the pregnant women at the beginning of the study.
  * The first interview will be face-to-face at the hospital.
  * A calendar will be created about home visits and timings for home midwifery care and counseling by meeting the pregnant woman at the hospital and obtaining their contact information.
  * Weekly home visits will be made to the pregnant women in the first month and training will be provided with the training booklet developed in line with the home midwifery care model based on the continuous midwifery care model during the home visits. Afterwards, two more home visits will be made to the pregnant women on a monthly basis and a total of 6 home visits will be made.
  * Pregnant women will be in constant communication via mobile phone.
  * After the sixth home visit, the Intention, Attitude and Behavior Scale in Gestational Diabetes and the Diabetes Self-Care Activities Questionnaire will be filled.
  Interventions: Other: Education
- Control (No Intervention): * All forms will be filled in by the pregnant women at the beginning of the study.
  * Pregnant women in the control group will not be subjected to any application other than the routine pregnancy follow-up and examinations recommended in the hospital.
  * Forms will be filled in parallel with the intervention group

INTERVENTIONS:
Other: Education — The training module, which will be developed in line with the continuous midwifery care model, will include home care and counseling of pregnant women with gestational diabetes (glucose monitoring and control, diet, exercise, evaluation of fetal health, etc.).
  Arms: Experimental

SUMMARY:
Since gestational diabetes carries the risk of serious complications for the mother and fetus, it is very important to follow up the pregnancy carefully and consciously. Home follow-up and prenatal care of these pregnant women, whose outpatient follow-up is continued without hospitalization, gains great importance. This study was planned as a randomized controlled experimental study to determine the effects of home midwifery care based on the continuous midwifery care model for pregnant women diagnosed with gestational diabetes, on the attitudes and self-care of pregnant women. The universe of this research, which will be carried out in a randomized controlled experimental type, will consist of pregnant women who applied to Çukurova University Balcalı Hospital Health Application and Research Center Gynecology and Obstetrics Department Pregnancy Polyclinic. The sample number was calculated by the Sample Size Calculator analysis and it was planned to include 24 participants in the experimental group and 24 participants in the control group. Single-blind randomized assignment and block randomization will be performed to avoid selection bias. The research will be conducted in the form of pre-test and post-test. The pre-test will be applied at the first encounter before the midwifery training, and the post-test will be applied after the 6th training. Data; It will be collected with the Pregnant Introductory Form, Intention, Attitude and Behavior Scale in Gestational Diabetes and Diabetes Self-Care Activities Questionnaire. Statistical Program for Social Science 22 will be used in data analysis. The data will be analyzed with appropriate analysis methods after testing for normality. The main subject of this research is to improve maternal and fetal health by providing continuous midwifery care at home for pregnant women who are diagnosed with gestational diabetes and are in the risky pregnancies group. With individual and continuous midwifery care provided at home, the self-care of women is strengthened and the intention, behavior and attitude towards both pregnancy and the health problem she has experienced are positively affected, contributing to the reduction of possible complications and providing a cost-effective service reveals the importance and necessity of the research.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled study to determine the effect of home midwifery care given to pregnant women diagnosed with gestational diabetes on the attitudes and self-care of pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Knowing Turkish and being literate
* Absence of fetal anomaly
* Having been diagnosed with gestational diabetes
* 24-28 and above gestational weeks

Exclusion Criteria:

* Communication difficulties

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnancy
Enrollment: 48 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Intention, Attitude and Behavior Scale in Gestational Diabetes | pre-intervention, immediately after the intervention, after 1 month. An increase in the score is interpreted as an increase in the level of knowledge and attitude about perinatal mental
  Change from the level of knowledge and awareness about perinatal mental health at 3 months
Diabetes Self-Care Activities Questionnaire | pre-intervention, immediately after the intervention, after 1 month. An increase in the score is interpreted as an increase in the level of knowledge and self care about perinatal mental
  Change from the level of knowledge and awareness about perinatal mental health at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cemile Onat Koroglu, Msc, Principal Investigator — Cukurova University
Locations (2):
- Turkey (Türkiye) (2):
  - Cemile Onat Koroglu, Adana
  - Cukurova University, Adana

IPD SHARING:
Plan to Share IPD: No